CLINICAL TRIAL: NCT02654327
Title: pRotective vEntilation With Veno-venouS Lung assisT in Respiratory Failure
Acronym: REST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); Northern Ireland Clinical Trials Unit (Other)
Responsible Party: Principal Investigator, Professor Danny McAuley, Professor of Intensive Care Medicine, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15084DMcA-AS; 13/143/02 (Other Grant/Funding Number: NIHR HTA)
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Failure With Hypoxia
Keywords: Extracorporeal; Acute Respiratory Distress Syndrome; Protective Lung Ventilation; Ventilator Induced Lung Injury; Carbon Dioxide Removal; Lung; Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Standard care with conventional lung protective mechanical ventilation
- ECCO2R to enable lower tidal volume mechanical ventilation (Experimental): VV-ECCO2R to enable lower tidal volume mechanical ventilation (target tidal volume of ≤ 3ml/kg predicted body weight and a Pplat ≤ 25cmH20)
  Interventions: Device: VV-ECCO2R to enable lower tidal volume mechanical ventilation

INTERVENTIONS:
Device: VV-ECCO2R to enable lower tidal volume mechanical ventilation — In the intervention arm a dual lumen catheter will be inserted into a central vein. VV-ECCO2R is commenced and managed as per study manual. Tidal volumes are then reduced on mechanical ventilation to enable lower tidal volume ventilation. Lower tidal volume facilitated by VV-ECCO2R will continue for a least 2 days up to a maximum of 7 days
  Arms: ECCO2R to enable lower tidal volume mechanical ventilation

SUMMARY:
This is a trial of a new way of treating patients with respiratory failure. The investigators propose to deliver a multi-centre clinical trial to determine whether veno-venous extracorporeal carbon dioxide removal (VV-ECCO2R) and lower tidal volume mechanical ventilation improves outcomes and is cost-effective, in comparison with standard care in patients who are mechanically ventilated for acute hypoxaemic respiratory failure

DETAILED DESCRIPTION:
Acute hypoxaemic respiratory failure requiring mechanical ventilation is a major cause of morbidity and mortality. A significant proportion of affected patients will have the Acute Respiratory Distress Syndrome (ARDS). Mechanical ventilation is often required to provide adequate gas exchange and although it is life-saving in this setting, it is also now known to contribute to the morbidity and mortality in the condition. Ventilators delivering high pressures and volumes cause regional over distension in the injured lung resulting in further inflammation and non-cardiogenic pulmonary oedema. The release of inflammatory mediators from the damaged lung causes systemic inflammation leading to multi-organ failure and death.

The few interventions that have been shown to reduce the high mortality in these patients have targeted ventilator-induced lung injury (VILI). A landmark trial by the ARDSNet trials group found that ventilating patients with acute hypoxaemic respiratory failure secondary to ARDS with a lung protective strategy aiming for a reduced tidal volume of 6ml/kg predicted body weight (PBW) and a maximum end-inspiratory plateau pressure (Pplat) ≤ 30cmH2O decreased mortality from 40% (in the conventional arm treated with tidal volume less than 12ml/kg PBW) to 31%.

Extracorporeal carbon dioxide removal (ECCO2R) in association with mechanical ventilation offers a potentially attractive solution to permit tidal volume reduction to less than 6ml/kg PBW and to achieve low plateau pressures (< 25cmH2O). Using these extracorporeal circuits, carbon dioxide can be 'dialysed' out of the blood while the lungs are ventilated in a more protective manner. In recent years, more efficient veno-venous devices have become available. These have replaced arterio-venous devices and have the advantage of not requiring arterial puncture. These can achieve carbon dioxide removal with relatively low extracorporeal blood flows (0.4-1 l/min) requiring only a smaller dual lumen venous catheter. In addition these ECCO2R devices use more biocompatible materials making the device more resistant to clot formation and cause less platelet and clotting factor consumption. Therefore only minimal systemic anticoagulation is required which reduces the likelihood of bleeding complications. These devices are now comparable to renal dialysis equipment, which is routinely used safely as standard care in ICUs in the United Kingdom.

Together this highlights the need for a large randomised controlled trial to establish whether VV-ECCO2R in acute hypoxaemic respiratory failure can allow the use of a more protective ventilatory strategy and is associated with improved patient outcomes. Importantly, if there was no benefit, the trial would provide evidence to stop the widespread adoption of an expensive and ineffective or potentially harmful treatment in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation using positive end expiratory pressure (PEEP) ≥ 5cmH2O
* Acute and potentially reversible cause of acute respiratory failure as determined by the treating physician
* Within 48 hours of the onset of hypoxemia as defined by Pa02/Fi02 less than or equal to 20kPA

Exclusion Criteria:

* Age < 16 years old
* Intubated and mechanically ventilated via an endotracheal or tracheostomy tube ≥ 7 days (168 hours) up to the time of randomisation
* Ability to maintain Vt to ≤ 3ml/kg PBW while maintaining pH ≥ 7.2 as determined by the treating physician
* Receiving, or decision to commence, ECMO in the next 24 hours
* Mechanical ventilation using high frequency oscillation ventilation or airway pressure release ventilation
* Untreated pulmonary embolism, pleural effusion or pneumothorax as the primary cause of acute respiratory failure
* Acute respiratory failure fully explained by left ventricular failure or fluid overload (May be determined by clinical assessment or echocardiography/cardiac output monitoring)
* Left ventricular failure requiring mechanical support
* Contra-indication to limited systemic anticoagulation with heparin
* Unable to obtain vascular access to a central vein (internal jugular or femoral vein)
* Consent declined
* Treatment withdrawal imminent within 24 hours
* Patients not expected to survive 90 days on basis of premorbid health status
* DNAR (Do Not Attempt Resuscitation) order (excluding advance directives) in place
* Severe chronic respiratory disease requiring domiciliary ventilation (except for sleep disordered breathing)
* Severe chronic liver disease (Child Pugh >11)
* Platelet count < 40,000 mm3 (Prior to catheter insertion)
* Previously enrolled in the REST trial
* Prisoners

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2016-05-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 90 days after randomisation

SECONDARY OUTCOMES:
Tidal volume (ml/kg Predicted Body Weight) | day 2 and day 3 after randomisation
Ventilator free days | 28 days after randomisation
Duration of ventilation in survivors | 28 days after randomisation
Need for Extracorporeal Membrane Oxygenation (ECMO) | 7 days after randomisation
Mortality rate | 28 days, 6 months and 1 year after randomisation
Health Related Quality of Life | 6 months and 1 year after randomisation
Adverse Event Rate | 28 days
Health & Social Care Service costs | 6 months and 1 year after randomisation
St George Respiratory Questionnaire | 1 year after randomisation
Need for home oxygen | 6 months and 1 year after randomisation
Post Traumatic Stress Syndrome Questionnaire (PTSS-14) | 1 year after randomisation
Montreal Cognitive Assessment (MoCA-BLIND) or AD8 Dementia Screening Interview (AD8) | 1 year after randomisation

OTHER OUTCOMES:
Right Ventricular function | Baseline & Day 2/Day 3
  Change in tricuspid annular plane systolic excursion (TAPSE) in cm at day 2 or 3 from randomisation measured with echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Fitzgerald M, Millar J, Blackwood B, Davies A, Brett SJ, McAuley DF, McNamee JJ. Extracorporeal carbon dioxide removal for patients with acute respiratory failure secondary to the acute respiratory distress syndrome: a systematic review. Crit Care. 2014 May 15;18(3):222. doi: 10.1186/cc13875. PMID 25033302
- [Background] Terragni PP, Del Sorbo L, Mascia L, Urbino R, Martin EL, Birocco A, Faggiano C, Quintel M, Gattinoni L, Ranieri VM. Tidal volume lower than 6 ml/kg enhances lung protection: role of extracorporeal carbon dioxide removal. Anesthesiology. 2009 Oct;111(4):826-35. doi: 10.1097/ALN.0b013e3181b764d2. PMID 19741487
- [Background] Bein T, Weber-Carstens S, Goldmann A, Muller T, Staudinger T, Brederlau J, Muellenbach R, Dembinski R, Graf BM, Wewalka M, Philipp A, Wernecke KD, Lubnow M, Slutsky AS. Lower tidal volume strategy ( approximately 3 ml/kg) combined with extracorporeal CO2 removal versus 'conventional' protective ventilation (6 ml/kg) in severe ARDS: the prospective randomized Xtravent-study. Intensive Care Med. 2013 May;39(5):847-56. doi: 10.1007/s00134-012-2787-6. Epub 2013 Jan 10. PMID 23306584
- [Derived] Boyle AJ, Reddy K, Conlon J, Auzinger G, Bannard-Smith J, Barrett NA, Camporota L, Gillies MA, Jackson C, McDowell C, Patel B, Perkins GD, Szakmany T, Tunnicliffe W, Welters ID, McNamee JJ, McAuley DF, O'Kane CM. Evaluation of Plasma Biomarkers to Understand the Biology and Heterogeneity of Treatment Effect in Lower Tidal Volume Ventilation Facilitated by Extracorporeal CO2 Removal in Acute Hypoxemic Respiratory Failure: A Secondary Analysis of the REST Trial. Crit Care Explor. 2025 Mar 27;7(4):e1246. doi: 10.1097/CCE.0000000000001246. eCollection 2025 Apr 1. PMID 40146037
- [Derived] Agus A, McNamee JJ, Jackson C, McAuley DF. Extracorporeal carbon dioxide removal compared to ventilation alone in patients with acute hypoxaemic respiratory failure: cost-utility analysis of the REST RCT. Health Technol Assess. 2023 Aug;29(33):1-34. doi: 10.3310/FCDQ8036. PMID 37843629
- [Derived] Boyle AJ, McDowell C, Agus A, Logan D, Stewart JD, Jackson C, Mills J, McNamee JJ, McAuley DF. Acute hypoxaemic respiratory failure after treatment with lower tidal volume ventilation facilitated by extracorporeal carbon dioxide removal: long-term outcomes from the REST randomised trial. Thorax. 2023 Aug;78(8):767-774. doi: 10.1136/thorax-2022-218874. Epub 2022 Oct 5. PMID 36198573
- [Derived] McNamee JJ, Gillies MA, Barrett NA, Perkins GD, Tunnicliffe W, Young D, Bentley A, Harrison DA, Brodie D, Boyle AJ, Millar JE, Szakmany T, Bannard-Smith J, Tully RP, Agus A, McDowell C, Jackson C, McAuley DF; REST Investigators. Effect of Lower Tidal Volume Ventilation Facilitated by Extracorporeal Carbon Dioxide Removal vs Standard Care Ventilation on 90-Day Mortality in Patients With Acute Hypoxemic Respiratory Failure: The REST Randomized Clinical Trial. JAMA. 2021 Sep 21;326(11):1013-1023. doi: 10.1001/jama.2021.13374. PMID 34463700
- [Derived] Stokes JW, Gannon WD, Rice TW. Extracorporeal Carbon Dioxide Removal or Extracorporeal Membrane Oxygenation: Why Should We Care? Crit Care Med. 2021 May 1;49(5):e546-e547. doi: 10.1097/CCM.0000000000004844. No abstract available. PMID 33854019

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02654327/SAP_000.pdf